CLINICAL TRIAL: NCT07308756
Title: Impact of Perioperative Dexmedetomidine and Esketamine on Postoperative Quality of Recovery in Patients Undergoing General Anesthesia and Surgery: A 2×2 Factorial Randomized Trial
Brief Title: Impact of Perioperative Dexmedetomidine and Esketamine on Postoperative Quality of Recovery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anaesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-0455
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: General Anesthesia; Surgery; Dexmedetomidine; Esketamine; Quality of Recovery
Keywords: General anesthesia; Surgery; Dexmedetomidine; Esketamine; Quality of recovery
MeSH Terms: interventions — Dexmedetomidine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine (Experimental): A loading dose of dexmedetomidine (0.2 ug/kg) is administered after anesthesia induction, followed by a continuous infusion of dexmedetomidineat a rate of 0.2 ug/kg/h until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with dexmedetomidine 100 ug and sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Interventions: Drug: Dexmedetomidine
- Esketamine (Experimental): A loading dose of esketamine (0.1 mg/kg) is administered after anesthesia induction, followed by a continuous infusion of esketamineat a rate of 0.1 mg/kg/h until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with esketamine 50 mg and sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Interventions: Drug: Esketamine
- Dexmedetomidine-esketamine (Experimental): A loading dose of dexmedetomidine (0.2 ug/kg) and esketamine (0.1 mg/kg) is administered after anesthesia induction, followed by a continuous infusion of dexmedetomidine at a rate of 0.2 ug/kg/h and esketamine at a rate of 0.1 mg/kg/h until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with dexmedetomidine 100 ug, esketamine 50 mg, and sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Interventions: Drug: Dexmedetomidine-esketamine
- Control (Placebo Comparator): A loading dose of placebo (normal saline) is administered after anesthesia induction, followed by a continuous infusion of placebo at a rate same as above until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — A loading dose of dexmedetomidine (0.2 ug/kg) is administered after anesthesia induction, followed by a continuous infusion of dexmedetomidineat a rate of 0.2 ug/kg/h until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with dexmedetomidine 100 ug and sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Arms: Dexmedetomidine
Drug: Esketamine — A loading dose of esketamine (0.1 mg/kg) is administered after anesthesia induction, followed by a continuous infusion of esketamineat a rate of 0.1 mg/kg/h until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with esketamine 50 mg and sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Arms: Esketamine
Drug: Dexmedetomidine-esketamine — A loading dose of dexmedetomidine (0.2 ug/kg) and esketamine (0.1 mg/kg) is administered after anesthesia induction, followed by a continuous infusion of dexmedetomidine at a rate of 0.2 ug/kg/h and esketamine at a rate of 0.1 mg/kg/h until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with dexmedetomidine 100 ug, esketamine 50 mg, and sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Arms: Dexmedetomidine-esketamine
Drug: Placebo — A loading dose of placebo (normal saline) is administered after anesthesia induction, followed by a continuous infusion of placebo at a rate same as above until 30 minutes before the end of surgery.
  Self-controlled analgesia is established with sufentanil 100 ug, diluated with normal saline to 100 ml, and programmed to deliver 2-ml boluses with a lock-out interval of 10 minutes and a background infusion rate at 1 ml/h for a duration of 48 hours.
  Arms: Control

SUMMARY:
For patients after surgery, quality of recovery has significant impacts on the prognosis, quality of life, and rational allocation of medical resources. Dexmedetomidine and esketamine have each been used during the perioperative period and improved postoperative analgesia and subjective sleep quality. This 2x2 factorial trial is designed to explore the effects of dexmedetomidine, esketamine, and their combination on the quality of recovery in patients recovering from surgery under general anesthesia.

DETAILED DESCRIPTION:
Surgical operation is an important therapeutic modality for surgical patients; quality of postoperative recovery has significant impacts on the prognosis, quality of life, and rational allocation of medical resources. Postoperative recovery is a complex process involving return of patients from surgery to baseline physiological and psychological status. Traditional indicators evaluating postoperative recovery mainly focus on physiological markers, length of hospital stay (LOS), and incidences of adverse events and complications. Recently, the quality of recovery (QoR) is increasingly used. QoR is subjectively reported by patients and includes multidimensional assessments on postoperative pain, cognitive function, sleep quality, and emotional stability.

Dexmedetomidine, a highly selective α2-adrenergic receptor agonist, has anxiolytic, sedative, and analgesic effects. By activing α2-adrenergic receptors in the locus coeruleus, it activates the endogenous sleep pathways, and produce a state mimicking non-rapid eye movement (NREM) sleep. Clinical studies showed that perioperative use of low-dose dexmedetomidine improves sleep architecture, increases sleep efficiency, and prolongs total sleep time in non-mechanically ventilated patients. Furthermore, when used as an analgesic adjuvant, dexmedetomidine improves analgesia, reduces opioid consumption, and reduces opioid-related adverse events.

Ketamine, a non-competitive N-Methyl-D-aspartic (NMDA) receptor antagonist, exerts analgesic and anti-hyperalgesic effects by reducing transmission of noxious stimuli to the spinal cord. It is characterized by minimal respiratory and circulatory depression and excellent analgesic efficacy. In recent years, multiple studies confirmed that ketamine has antidepressant properties. Ketamine is a racemic mixture composed of S-ketamine (esketamine) and R-ketamine. Esketamine exhibits a stronger affinity for the NMDA receptor, with an effect approximately twice that of racemic ketamine. In clinical practice, esketamine has stronger analgesic effects and a lower incidence of adverse psychomimetic reactions. When used in combination with opioids, esketamine improved postoperative analgesia.

Previous studies showed that combined use of dexmedetomidine and esketamine might produce synergetic effects in improving sedation and analgesia. A recent trial found that low-dose dexmedetomidine-esketamine combination improved pain relief and subjective sleep quality in patients after scoliosis corrective surgery, without increasing side effects. It is therefore hypothesized that co-administration of dexmedetomidine and esketamine may enhance efficacy and optimize the quality of postoperative recovery. This 2x2 factorial trial is designed to explore the effects of dexmedetomidine, esketamine, and their combination on the quality of recovery in patients recovering from surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over;
* Scheduled to undergo surgery under general anesthesia, with an expected surgical duration of at least 1 hour;
* Required patient-controlled intravenous analgesia after surgery.

Exclusion Criteria:

* Unable to communicate preoperatively due to visual, auditory, or verbal barriers or other reasons;
* Severe bradycardia (heart rate <50 bpm), sick sinus syndrome, or grade 2 or higher atrioventricular block without pacemaker;
* History of hyperthyroidism or pheochromocytoma;
* History of schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis, or intracranial hypertension;
* Intracranial tumor or neurosurgery;
* Severe liver dysfunction (Child-Pugh class C), renal failure (requiring renal replacement therapy), or American Society of Anesthesiologists class IV or higher;
* Enrolled in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery-15 (QoR-15) score | At 24 hours after surgery
  A 15-item scale that evaluate quality of recovery in five dimensions: pain, physiological comfort, physiological independence, psychological support, and emotional state. Scores range from 0 to 150 , with higher scores indicating better recovery quality.

SECONDARY OUTCOMES:
Quality of recovery-15 (QoR-15) score | At 72 hours after surgery
  QoR is a 15-item scale that evaluate quality of recovery in five dimensions: pain, physiological comfort, physiological independence, psychological support, and emotional state. Scores range from 0 to 150 , with higher scores indicating better recovery quality.
Postoperative delirium (POD) within 4 days | Up to 4 days after surgery
  Delirium will be assessed twice daily (8:00-10:00 and 18:00-20:00) using the 3-minute diagnostic interview for confusion assessment method-defined delirium (3D-CAM) or the confusion assessment method for the intensive care unit (CAM-ICU).
Incidence of delayed neurocognitive recovery at 5 days | Up to 5 days after surgery
  Cognitive function will be assessed with the telephone-administered Montreal Cognitive Assessment (T-MoCA) at baseline and at 5 days or before hospital discharge after surgery. A decline of T-MoCA score of 1 standard deviation (SD) or more from baseline is defined as delayed neurocognitive recovery.

OTHER OUTCOMES:
Area under curve of pain intensity after surgery | Up to 4 days after surgery
  Pain intensity will be assessed at 1 hour and then twice daily (8:00-10:00 and 18:00-20:00) after surgery using the numeric rating scale (an 11-point scale where 0=no pain and 10=the worst pain).
Cumulative subjective sleep quality score after surgery | Up to 4 days after surgery
  Subjective sleep quality will be assessed once daily (8:00-10:00) after surgery using the numeric rating scale (an 11-point scale where 0=the best sleep and 10=the worst sleep).
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery.
Incidence of postoperative complications within 30 days | Up to 30 days after surgery
  Postoperative complications are generally defined as new-onset medical conditions that are deemed harmful and required therapeutic intervention, i.e., grade 2 or higher on the Clavien-Dindo classification.
All-cause 30-day mortality | Up to 30 days after surgery
  All-cause 30-day mortality
Incidence of delayed neurocognitive recovery at 30 days | At 30 days after surgery
  Cognitive function will be assessed with the telephone-administered Montreal Cognitive Assessment (T-MoCA) at baseline and at 30 days after surgery. A decline of T-MoCA score of 1 standard deviation (SD) or more from baseline is defined as delayed neurocognitive recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Background] Guo J, Qiu D, Gu HW, Wang XM, Hashimoto K, Zhang GF, Yang JJ. Efficacy and safety of perioperative application of ketamine on postoperative depression: A meta-analysis of randomized controlled studies. Mol Psychiatry. 2023 Jun;28(6):2266-2276. doi: 10.1038/s41380-023-01945-z. Epub 2023 Jan 20. PMID 36670198
- [Background] Xie M, Liang Y, Deng Y, Li T. Effect of S-ketamine on Postoperative Pain in Adults Post-Abdominal Surgery: A Systematic Review and Meta-analysis. Pain Physician. 2023 Jul;26(4):327-335. PMID 37535771
- [Background] Wang S, Deng CM, Zeng Y, Chen XZ, Li AY, Feng SW, Xu LL, Chen L, Yuan HM, Hu H, Yang T, Han T, Zhang HY, Jiang M, Sun XY, Guo HN, Sessler DI, Wang DX. Efficacy of a single low dose of esketamine after childbirth for mothers with symptoms of prenatal depression: randomised clinical trial. BMJ. 2024 Apr 10;385:e078218. doi: 10.1136/bmj-2023-078218. PMID 38808490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Focus (Am Psychiatr Publ). 2019 Jan;17(1):55-65. doi: 10.1176/appi.focus.17105. Epub 2019 Jan 7. PMID 32015715
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Smith-Apeldoorn SY, Veraart JK, Spijker J, Kamphuis J, Schoevers RA. Maintenance ketamine treatment for depression: a systematic review of efficacy, safety, and tolerability. Lancet Psychiatry. 2022 Nov;9(11):907-921. doi: 10.1016/S2215-0366(22)00317-0. PMID 36244360
- [Background] Ma S, Chen M, Jiang Y, Xiang X, Wang S, Wu Z, Li S, Cui Y, Wang J, Zhu Y, Zhang Y, Ma H, Duan S, Li H, Yang Y, Lingle CJ, Hu H. Sustained antidepressant effect of ketamine through NMDAR trapping in the LHb. Nature. 2023 Oct;622(7984):802-809. doi: 10.1038/s41586-023-06624-1. Epub 2023 Oct 18. PMID 37853123
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Lu W, Fu Q, Luo X, Fu S, Hu K. Effects of dexmedetomidine on sleep quality of patients after surgery without mechanical ventilation in ICU. Medicine (Baltimore). 2017 Jun;96(23):e7081. doi: 10.1097/MD.0000000000007081. PMID 28591048
- [Background] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372
- [Background] Tasbihgou SR, Barends CRM, Absalom AR. The role of dexmedetomidine in neurosurgery. Best Pract Res Clin Anaesthesiol. 2021 Jul;35(2):221-229. doi: 10.1016/j.bpa.2020.10.002. Epub 2020 Oct 14. PMID 34030806
- [Background] Mo Y, Zimmermann AE. Role of dexmedetomidine for the prevention and treatment of delirium in intensive care unit patients. Ann Pharmacother. 2013 Jun;47(6):869-76. doi: 10.1345/aph.1AR708. PMID 23719785
- [Background] Xu M, Zhang G, Tang Y, Wang R, Yang J. Impact of Regional Anesthesia on Subjective Quality of Recovery in Patients Undergoing Thoracic Surgery: A Systematic Review and Meta-Analysis. J Cardiothorac Vasc Anesth. 2023 Sep;37(9):1744-1750. doi: 10.1053/j.jvca.2023.05.003. Epub 2023 May 5. PMID 37301699
- [Background] Joe YE, Kang CM, Lee HM, Kim KJ, Hwang HK, Lee JR. Quality of Recovery of Patients Who Underwent Curative Pancreatectomy: Comparison of Total Intravenous Anesthesia Versus Inhalation Anesthesia Using the QOR-40 Questionnaire. World J Surg. 2021 Aug;45(8):2581-2590. doi: 10.1007/s00268-021-06117-0. Epub 2021 Apr 21. PMID 33881579
- [Background] Hung KC, Ko CC, Hsu CW, Pang YL, Chen JY, Sun CK. Association of peripheral nerve blocks with patient-reported quality of recovery in female patients receiving breast cancer surgery: a systematic review and meta-analysis of randomized controlled studies. Can J Anaesth. 2022 Oct;69(10):1288-1299. doi: 10.1007/s12630-022-02295-0. Epub 2022 Jul 26. PMID 35882724
- [Background] Hung KC, Chu CC, Hsing CH, Chang YP, Li YY, Liu WC, Chen IW, Chen JY, Sun CK. Association between perioperative intravenous lidocaine and subjective quality of recovery: A meta-analysis of randomized controlled trials. J Clin Anesth. 2021 Dec;75:110521. doi: 10.1016/j.jclinane.2021.110521. Epub 2021 Sep 20. PMID 34547603
- [Background] Nilsson U, Gruen R, Myles PS. Postoperative recovery: the importance of the team. Anaesthesia. 2020 Jan;75 Suppl 1:e158-e164. doi: 10.1111/anae.14869. PMID 31903575
- [Background] Campfort M, Cayla C, Lasocki S, Rineau E, Leger M. Early quality of recovery according to QoR-15 score is associated with one-month postoperative complications after elective surgery. J Clin Anesth. 2022 Jun;78:110638. doi: 10.1016/j.jclinane.2021.110638. Epub 2022 Jan 13. PMID 35033845
- [Background] Shulman MA, Myles PS, Chan MT, McIlroy DR, Wallace S, Ponsford J. Measurement of disability-free survival after surgery. Anesthesiology. 2015 Mar;122(3):524-36. doi: 10.1097/ALN.0000000000000586. PMID 25689757
- [Background] Tahiri M, Sikder T, Maimon G, Teasdale D, Hamadani F, Sourial N, Feldman LS, Guralnick J, Fraser SA, Demyttenaere S, Bergman S. The impact of postoperative complications on the recovery of elderly surgical patients. Surg Endosc. 2016 May;30(5):1762-70. doi: 10.1007/s00464-015-4440-2. Epub 2015 Jul 21. PMID 26194260